CLINICAL TRIAL: NCT03531190
Title: A Randomized Controlled Clinical Trial of Pre- and Postoperative Supplementation With Zinc, Vitamin C, Arginine and Multivitamin Mineral in Patients Treated for Head and Neck Cancer
Brief Title: Pre- and Postoperative Nutrition in Head and Neck Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jens Rikardt Andersen, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-17040654
Record Dates: First submitted 2018-04-09; First posted 2018-05-21 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Head and Neck Cancer
Keywords: Head and neck cancer; wound healing; pre and post-surgical nutrition; zinc, arginine, vitamin C, protein, oral supplements
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Dietary Supplements; Proteins

STUDY DESIGN:
Intervention Model Description: Randomized to intervention. Control is the present treatment in the department + protein supplementation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional supplement (Protein + MIX) (Experimental): Patients are given: Nutritional Supplement of protein 2-3 times a day + MIX once daily for 35 days
  Interventions: Dietary Supplement: Nutritional supplement (Protein + MIX)
- Nutritional supplement (Protein) (Active Comparator): Nutritional Supplement of protein as needed 2-3 times a day for 35 days
  Interventions: Dietary Supplement: Nutritional supplement (Protein)

INTERVENTIONS:
Dietary Supplement: Nutritional supplement (Protein + MIX) — Protein supplement as needed + 750 mg vitamin C, 15 g. arginine, 35 mg. zinc and two multivitamin tablets, by mouth every day for 35 days.
  Arms: Nutritional supplement (Protein + MIX)
Dietary Supplement: Nutritional supplement (Protein) — Protein supplement as needed
  Arms: Nutritional supplement (Protein)

SUMMARY:
The purpose of the project is to investigate the effect of wound healing of a combined pre- and postoperative oral supplement, consisting of zinc, vitamin C, arginine and multivitamin, as a supplement for adequate nutrition in patients operated for head and neck cancer.

DETAILED DESCRIPTION:
The project will be conducted as an open, randomized intervention study, and includes patients with head and neck cancer that are planned for operation. 40 participants are allocated to the intervention or control group, respectively. For both groups, the experiment will last for five to six weeks, depending on when the trial participants are planned for surgery. The intervention group must take a dietary supplement and a protein drink for 35 days (7 days preoperatively and 28 days postoperatively), which is delivered 7 days preoperatively. The same applies to the control group that only receives protein drinks. The length of the intervention period is based on the design of previous studies. During the project, compliance will be evaluated by counting the amount of remaining dietary supplements and protein drinks that the participants return on a regular basis. The control group receives standard treatment as well as protein drinks. For all participants included in the experiment blood tests and an ultrasound scanning will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Authorized/legal age (> 18 years)
* Patients who understand written and oral Danish, and are able to give written consent
* Patients diagnosed with head and neck cancer, which are set for surgery
* Patients operated on the outside of the neck

Exclusion Criteria:

* Patients who do not understand, speak or write Danish
* Not Authorized/not legal age (<18 years)
* Pregnant and breastfeeding women
* Patients previously employed in the field of surgery within the last 5 years (prior years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
POSAS-scale (The Patient and Observer Scar Assessment Scale v2.0 / EN) | 2 months
  points on POSAS-questionaire (7-70)

SECONDARY OUTCOMES:
Appearance of the scar (scale) | 2 months
  blind professional rating based on rank (from photographs)(1-10)
Ultrasound scanning | 2 months
  Number of cavities in the wound
Biochemical measurements (micromol/l) at start and finish | 2 months
  Changes in the concentrations of micronutrients in the intervention period:
  p-albumin, p-C-Reactive Protein, p-cobalamin, p-folic acid, p-magnesium, p-ferritin
Size of the scar (cm) | 2 months
  measured with ruler

OTHER OUTCOMES:
Peripheral oxygen tension (partial pressure, kPa) | 2 months
  Peripheral oxygen tension measured on the finger tip
Difficulty in swallowing (scale) | 2 months
  assessed by rank-scale (1-100)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Rikardt R Andersen, MD,MPA, Principal Investigator — University of Copenhagen, Department of Nutrition, Exercise and Sports
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No